CLINICAL TRIAL: NCT05022654
Title: Phase II Clinical Study to Evaluate the Efficacy and Safety of SI-B001 Combined With Irinotecan in the Treatment of Recurrent and Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: SI-B001 Combined With Irinotecan in the Treatment of Recurrent Metastatic Esophageal Squamous Cell Carcinoma.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SI-B001_207
Record Dates: First submitted 2021-08-22; First posted 2021-08-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Squamous Cell Carcinomas
Keywords: ESCC
MeSH Terms: interventions — Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SI-B001 combined with irinotecan (Experimental): Patients with recurrent metastatic esophageal squamous cell carcinoma who had failed first-line therapy with PD-1(L1) monoclonal antibody plus platinum-based chemotherapy were enrolled.
  Interventions: Drug: SI-B001; Drug: Irinotecan

INTERVENTIONS:
Drug: SI-B001 — Administered by intravenous drip every 2 weeks (Q2W). The first intravenous infusion is 120 min±10min. If the infusion reaction can be tolerated during the first infusion, the subsequent infusion can be completed in 60-120 min.
Drug: Irinotecan — The dose of irinotecan was 180mg/m2 Q2W, the infusion method was according to the drug instructions, SI-B001 and irinotecan were used on the same day, and irinotecan was injected after SI-B001 infusion.

SUMMARY:
This multi-center, open label Phase II clinical study is performed in patients with relapsed and metastatic esophageal squamous cell carcinoma progressed on prior PD-1/L1 antibody with or without chemotherapy. This study is investigating the safety and efficacy of SI-B001 at optimal combination dose with irinotecan in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. Male or female, age: ≥18 years and ≤75 years;
3. Expected survival time ≥3 months;
4. Locally advanced esophageal squamous cell carcinoma confirmed histologically or pathologically as recurrent or metastatic or without indications of radical local treatment;
5. Patients who failed or were intolerant to first-line anti-PD-1 (L1) monoclonal antibody plus platinum-based chemotherapy
6. Agree to provide archived tumor tissue specimens of primary or metastatic lesion (4 surgical specimens (thickness 5μm) without staining section (anti-removal);6 unstained sections (anti-removal) surgical specimens (thickness 10μm) or fresh tissue samples, if the patient cannot provide, can be included after the investigator's judgment;
7. There must be at least one measurable lesion conforming to the RECIST V1.1 definition. Tumor lesion located in the area of previous radiotherapy or other local and regional treatment sites is generally not a measurable lesion unless there is definite progression of the lesion or the lesion persists three months after radiotherapy;
8. Physical fitness ECOG score of 0 or 1;
9. Toxicity from previous antitumor therapy has returned to ≤1 as defined by NCI-CTCAE V5.0 (except for toxicity that the investigators determined to be of no safety risk, such as hair loss, grade 2 peripheral neurotoxicity, and stabilized hypothyroidism after hormone replacement therapy);
10. Organ function levels must meet the following requirements and meet the following standards:

    A) Bone marrow function: absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet count ≥90×10^9/L, hemoglobin ≥90 g/L; B) Liver function: Total bilirubin TBIL≤1.5×ULN (total bilirubin ≤3×ULN in Subjects with Gilbert's syndrome, liver cancer or liver metastasis), AST and ALT ≤2.5×ULN in patients without liver metastasis, AST and ALT ≤5.0×ULN in patients with liver metastasis; C) Renal function: Creatinine (Cr) ≤1.5×ULN, or creatinine clearance (Ccr) ≥50 mL/min (according to Cockcroft and Gault formula); D) Urine routine / 24-hour protein quantification: qualitative urine protein ≤1+ (if qualitative urine protein ≥2+, 24 hours < 1g can be included); E) Cardiac function: left ventricular ejection fraction ≥50%; F) Coagulation function: International standardized ratio (INR) ≤1.5×ULN, and activated partial thrombin time (APTT) ≤1.5×ULN;
11. Eligible patients (male and female) who are fertile must agree to use a reliable contraceptive method (hormonal or barrier method or abstinence, etc.) with their partner during the trial and for at least 6 months after the last medication;Women of childbearing age must have a negative blood or urine pregnancy test within 7 days prior to the first use of the study drug.

Exclusion Criteria:

1. Have received chemotherapy, radiotherapy, biotherapy, endocrine therapy, immunotherapy and other anti-tumor therapy within 4 weeks prior to the first use of the study drug, except for the following:

   Oral fluorouracil and small molecule targeted drugs were used within 2 weeks before the first administration of the study drug or within 5 half-lives of the drug; The traditional Chinese medicines with anti-tumor indications were within 2 weeks before the first use of the study drug;
2. Patients with esophageal fistula;
3. Received an unmarketed clinical investigational drug or treatment within 4 weeks prior to initial use of the investigational drug;
4. Had major organ surgery (excluding needle biopsy, tracheotomy, gastrostomy, etc.) or had significant trauma within 4 weeks prior to the first use of study drugs, or needed to undergo elective surgery during the trial;
5. Previous allogeneic hematopoietic stem cell transplantation or organ transplantation;
6. A history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

   Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, grade iii atrioventricular block, etc； In the resting state, QT interval was prolonged (QTc > 450 msec in men or QTc > 470 msec in women)； Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other grade 3 or higher cardio-cerebrovascular events within 6 months prior to the first administration; New York Heart Association (NYHA) heart function grade ≥II heart failure;
7. Active autoimmune and inflammatory diseases, such as systemic lupus erythematosus, inflammatory bowel disease, etc., except type I diabetes, hypothyroidism that can be controlled only with replacement therapy, and skin diseases that do not require systemic treatment;
8. Patients with a history of other malignant tumors and signs of recurrence and metastasis within 1 year before the first administration;
9. Poorly controlled hypertension (systolic blood pressure & GT;150 mmHg or diastolic pressure >100 mmHg);
10. Pulmonary disease of grade 3 or higher defined by CTCAE V5.0;Patients with past or present interstitial lung disease (ILD);
11. Cerebral parenchymal or meningeal metastases with clinical symptoms were not suitable for inclusion.
12. Previous use of anti-EGFR antibody drug therapy;
13. There are known allergic contraindications to any excipients of SI-B001 or irinotecan;
14. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection or hepatitis C virus infection;
15. Active infections requiring systemic treatment, such as severe pneumonia, bacteremia, septicemia, etc；'
16. Pregnant or lactating women;
17. Persons with mental disorders or poor compliance;
18. The investigator considers that the subject has a history of other serious systemic diseases or other reasons to be unsuitable for this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to approximately 24 months
  objective response rate
Optimal combination dose (only IIa) | Up to approximately 24 months
  Optimal combination dose of SI-B001 with irinotecan(only IIa)

SECONDARY OUTCOMES:
PFS | Up to approximately 24 months
  Progression-Free-Survival
DCR | Up to approximately 24 months
  Disease-control rate
DOR | Up to approximately 24 months
  Duration of Response
OS | Up to approximately 24 months
  Overall Survival
TEAE | Up to approximately 24 months
  Treatment Emergent Adverse Events
Cmax | Up to approximately 24 months
  Maximum serum concentration
Tmax | Up to approximately 24 months
  Time to maximum serum concentration
Ctrough | Up to approximately 24 months
  Minimum serum concentration
ADA | Up to approximately 24 months
  anti-SI-B001 antibody

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (6):
- China (6):
  - Beijing Cancer Hostital, Beijing, Beijing Municipality
  - Anyang Cancer Hospital of Henan Province, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Suining Central Hospital, Suining, Sichuan